CLINICAL TRIAL: NCT06945211
Title: Task Oriented Mirror Therapy for Upper Limb Motor Function in Stroke Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/65
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Stroke Patients
Keywords: Mirror Therapy; Stroke; Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP A LOW INTENSITY TASK ORIENTED MIRROR THERAPY (Experimental): Subjects will recieve Low Intensity Task Oriented Mirror Therapy:
  Mirror will be placed on table perpendicular to patient in such a way that the reflection of unaffected arm to be seen.
  The subject will be instructed to perform movement with unaffected arm. Task oriented activities: grasping objects, handling water cups, folding towels, spoon feeding, stacking wooden blocks.
  Interventions: Procedure: LOW INTENSITY TASK ORIENTED MIRROR THERAPY
- INTERVENTION GROUP B HIGH INTENSITY TASK ORIENTED MIRROR THERAP (Experimental): Subjects will receive High Intensity Task Oriented Mirror Therapy :
  Mirror will be placed on table perpendicular to patient in such a way that the reflection of unaffected arm to be seen.
  The subjects will be instructed to perform movement with unaffected arm. Task Oriented Activities: grasping objects, handling water cups, folding towels, spoon feeding, stacking wooden blocks.
  Interventions: Procedure: High Intensity Task Oriented Mirror Therapy

INTERVENTIONS:
Procedure: LOW INTENSITY TASK ORIENTED MIRROR THERAPY — Group A Low Intensity Task Oriented Mirror Therapy will be administered for 2 and half hour per week for 30 min a day, 10 rep five times a week for 8 weeks.
  Task-oriented Activities for Group A:
  Using Sponge Balls Reaching and Grasping Objects. Handling Water Cups(pouring water ) Wiping with Rags (cleaning a table ). Using a Spray Bottle Writing and Drawing Folding Towels Turning Pages Brushing Hair keyboard typing Grabbing and releasing a cup. Spoon Feeding Practice Drinking from a Cup Card flip activity Stacking Wooden Blocks Total number of sessions 40 , 5 days a week for 30 min with 10 reps per day for 8 consecutive weeks.
  Arms: INTERVENTION GROUP A LOW INTENSITY TASK ORIENTED MIRROR THERAPY
Procedure: High Intensity Task Oriented Mirror Therapy — Group B High Intensity Task Oriented Mirror Therapy will be administered for 5 hours per week for 60 min a day, 20 rep five times a week for 8 weeeks. The mode of mirror therapy will be unilateral as subjects will perform movement only on unaffected arm.
  Task-oriented Activities for Group B:
  Using Sponge Balls Reaching and Grasping Objects. Handling Water Cups(pouring water ) Wiping with Rags (cleaning a table ). Using a Spray Bottle Writing and Drawing Folding Towels Turning Pages Brushing Hair keyboard typing Grabbing and releasing a cup. Spoon Feeding Practice Drinking from a Cup Card flip activity Stacking Wooden Blocks Total number of sessions 40 , 5 days a week for 60 min with 20 reps per day for 8 consecutive weeks
  Arms: INTERVENTION GROUP B HIGH INTENSITY TASK ORIENTED MIRROR THERAP

SUMMARY:
Stroke remains a major public health disease worldwide ,it usually associating with damage to the motor function and other functional disabilities. Persistent upper extremity dysfunction affects many post strokepatients and is strongly associated with decreased activities of daily living . Mirror therapy one of the rehabilitation that is beneficial for neuroplasticity .This therapy is used to improve motor function after stroke .

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are :

1. To imorove upper limb motor function and
2. To improve activities of daily lving .
3. To enhance motor skills.

HYPOTHESIS:

Alternate Hypothesis:

There will be statisticallly significant difference in high intensity task oriented mirror therapy and low intensity task oriented mirror therapy on upper limb motor function ,activities of daily living and enhancing motor skills in stroke patients (p<0.05)

Null Hypothesis:

There will be no statisticallly significant difference in high intensity task oriented mirror therapy and low intensity task oriented mirror therapy on upper limb motor function

,activities of daily living and enhancing motor skills in stroke patients (p>0.05)

RESEARCH DESIGN : Experimental study .Randomized control trail.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age of patient 45 years and above
* Both ischemic and hemorrhagic stroke ( subacute and chronic stroke). Cognitive function relatively intact score > 24 MoCA
* The patient can sit with / without support for more than 30 min

Exclusion Criteria:

* Subjects with visual impairments or unilateral neglect.
* having global aphasia.
* unstable medical conditions or comorbidities.
* score 3 and above on modified ashworth scale.
* patient with orthopedic condition or any fractures.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
UPPER LIMB MOTOR FUNCTION | 10 weeks
  MOTOR FUNCTION WILL BE ASSESSED USING FUGL MEYER ASSESSMENT OF UPPER LIMB AS THE MAIN OUTCOME MEASURE .

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan